CLINICAL TRIAL: NCT02013323
Title: Clinical and Microbiological Efficacy of Systemic Ayurvedic Immunomodulator Septilin in the Treatment of Chronic Periodontitis-- A Randomized Controlled Clinical Trial.
Brief Title: Clinical and Microbiological Efficacy of Systemic Ayurvedic Immunomodulator Septilin in the Treatment of Chronic Periodontitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Government Dental College and Research Institute, Bangalore (Other)
Collaborators: Himalaya Drug Company Ltd. India (Unknown)
Responsible Party: Principal Investigator, Dr. A R Pradeep, Professor, Government Dental College and Research Institute, Bangalore
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GDCRI/ACM/PG/PhD/10/2013-14
Record Dates: First submitted 2013-12-08; First posted 2013-12-17 (Estimated); Last update posted 2013-12-17 (Estimated); Status verified 2013-12

CONDITIONS: Chronic Periodontitis
Keywords: Septiline, chronic periodontitis, Immunomodulator, microbiology
MeSH Terms: conditions — Chronic Periodontitis | interventions — Tooth Exfoliation; Root Planing; septilin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Septilin Group (Active Comparator): Subjects in septilin group received Septilin tablets (Septilin tablets, Himalaya Drug Company, India), 500 mg of 2 tablets to be taken thrice daily for 7 days after scaling and root planing
  Interventions: Drug: Scaling and root planing, and Septilin for 7 days
- Placebo Group (Placebo Comparator): Subjects in placebo group received Placebo tablets thrice daily for 7 days after Scaling and root planing
  Interventions: Drug: Scaling and root planing, and Placebo drug for 7 days

INTERVENTIONS:
Drug: Scaling and root planing, and Septilin for 7 days — Subjects in septilin group received Septilin tablets (Septilin tablets, Himalaya Drug Company, India), 500 mg of 2 tablets to be taken thrice daily for 7 days after scaling and root planing and checked for clinical and micrbiological parameters at baseline, 10 days, 1 month, 3 months and 6 months.
  Arms: Septilin Group
Drug: Scaling and root planing, and Placebo drug for 7 days — Subjects in placebo group received placebo tablets taken thrice daily for 7 days and checked for clinical and microbiological parameters at baseline, 10 days, 1 month, 3 months and 6 months
  Arms: Placebo Group

SUMMARY:
The present clinical trial was designed to investigate the clinical and microbiological effectiveness of systemic ayurvedic immunomodulator Septilin as an adjunct to scaling and root planing (SRP) in the treatment of chronic periodontitis (CP)

DETAILED DESCRIPTION:
OBJECTIVE: The present clinical trial was designed to investigate the clinical and microbiological effectiveness of systemic ayurvedic immunomodulator Septilin as an adjunct to scaling and root planing (SRP) in the treatment of chronic periodontitis (CP).

DESIGN: Sixty five subjects presenting at least twelve teeth with probing depth (PD) ≥4 mm were selected. 33 subjects were randomly assigned to full-mouth SRP + Septilin (group 1) and 32 subjects were assigned to full-mouth SRP + Placebo (group 2). The clinical outcomes evaluated were plaque index (PI), gingival index (GI), clinical attachment level (CAL), PD and % of sites with bleeding on probing (%BOP) at baseline (B\L), 10 days, 1, 3 and 6 months interval and percentage of sites positive for A. actinomycetemcomitans, P. gingivalis and T. forsythia were recorded at B/L, 3 and 6 months using polymerase chain reaction.

ELIGIBILITY:
Inclusion Criteria:

* age 30 to 50 years
* atleast 12 scorable teeth with a probing depth (PD) ≥ 4 mm not including third molars
* teeth with orthodontic appliances bridges, crowns, or implants
* radiographic evidence of bone loss.

Exclusion Criteria:

* pregnancy or lactation
* smokers
* systemic diseases like diabetes mellitus, immunocompromised patients
* systemic antibiotics taken within the previous 6 months
* use of non-steroidal anti-inflammatory drugs
* sub-gingival SRP or surgical periodontal therapy in the previous year.

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2013-03; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Clinical Attachment Level (CAL) | Gain in CAL from Baseline to 6 month
  The primary outcome of the study was gain in CAL from Baseline to 6 month

SECONDARY OUTCOMES:
PIaque Index (PI), Gingival Index (GI), Probing Depth (PD), % Bleeding on Probing and reduction in number of sites positive for each microbial species | The differences in PI, GI, PD, %BOP between two groups and reduction in number of sites positive for each microbial species from Baseline to 6 month
  The differences in PI, GI, PD, %BOP between two groups and reduction in number of sites positive for each microbial species from Baseline to 6 months

CONTACTS AND LOCATIONS:
Overall Officials: A R Pradeep, MDS, Principal Investigator — Govt Dental College and Research Institute
Locations (1):
- Government Dental College and Research Institute, Bangalore, Karnataka, India